## **Study Protocol**

Official Title: Determining the Impact of Creative Drama on Gender Role Stress, Attitudes Toward Violence Against Women, and Aggression Among Men Affected by the 2023 Earthquake in Türkiye

NCT Number: NCT Pending

Responsible Party: Dr. Aslı SİS ÇELİK, Principal Investigator, Atatürk University

Ethics Committee Approval: Approved by the Atatürk University Faculty of Medicine Non-Interventional Clinical Research Ethics Committee

Study Period: November 2025 – December 2026

## 1. Background and Rationale

Two major earthquakes (7.7 and 7.6 magnitudes) occurred in Türkiye on February 6, 2023, affecting 11 provinces, including Kahramanmaraş, Hatay, Adıyaman, and Malatya. These disasters caused not only physical destruction but also long-term psychological and social trauma among survivors. Research indicates that earthquakes can trigger high levels of stress, post-traumatic stress disorder, depression, aggression, and tendencies toward violence. Creative Drama, as a non-pharmacological and interactive psychosocial intervention, has been found to reduce stress and anxiety, improve empathy and communication, and promote social cohesion. This randomized controlled experimental study aims to determine the impact of Creative Drama on gender role stress, attitudes toward violence against women, and aggression in men who experienced the 2023 earthquake in Türkiye.

# 2. Objectives

Primary Objective: To evaluate the effect of Creative Drama on gender role stress, attitudes toward violence against women, and aggression among earthquake-affected men. Secondary Objectives: To explore potential improvements in empathy, communication skills, and psychological well-being following Creative Drama sessions.

## 3. Study Design

The study will use a randomized controlled experimental design with three parallel arms: (1) Experimental Group (Creative Drama Program), (2) Placebo Group (Film Viewing Sessions), (3) Control Group (No Intervention). Participants will be randomly assigned to one of the three groups using simple randomization generated through randomizer.org. The study will employ a double-blind design, where participants and the outcome assessor will be blinded to group assignments.

# 4. Participants and Sampling

The study population will consist of men residing in Malatya who experienced the February 6, 2023 earthquake. Participants will be recruited via social media announcements. The required sample size was determined using a G\*Power analysis, indicating 22 participants per group for a large effect size (0.80), a significance level of 0.05, and 90% power. To account for potential dropouts, 25 participants will be included in each group, for a total of 75 men.

### 5. Inclusion and Exclusion Criteria

Inclusion: Males aged 18–65 years, experienced the earthquake, married, volunteers, no disabilities or psychiatric diagnoses, no prior creative drama or psychosocial support, agree to attend sessions. Exclusion: Withdrawal, irregular attendance, relocation, divorce, or receiving psychosocial support during the study.

#### **6. Intervention Procedures**

Experimental Group: 10 weekly Creative Drama sessions (90 minutes each). Placebo Group: Watching 10 Turkish films (one per week) with themes of masculinity and violence. Control Group: No intervention; pretest and posttest only.

## 7. Data Collection Tools

Participant Information Form, Gender Role Stress Scale for Men, Attitudes Toward Violence Against Women Scale, Buss-Perry Aggression Questionnaire – Short Form.

## 8. Data Analysis Plan

Data will be analyzed using SPSS by an independent statistician blinded to group assignments (coded X, Y, Z). Analyses: descriptive stats, t-tests, ANOVA, repeated measures; significance p < 0.05.

## 9. Ethical Considerations

Approved by Atatürk University Faculty of Medicine Non-Interventional Clinical Research Ethics Committee. Written informed consent will be obtained from participants. Data will be stored securely and used only for research purposes.

### 10. Expected Outcomes

Creative Drama is expected to reduce gender role stress and aggression and improve attitudes toward women and emotional expression among men who experienced the earthquake.